CLINICAL TRIAL: NCT01202643
Title: G-CSF and Endometrial Growth, Embryo Implantation and Pregnancy Following FET or Donor ET
Brief Title: Effect of Colony Stimulating Factor on Poor Endometrial Development During IVF
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Center for Human Reproduction (Other)
Collaborators: Foundation for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, David H. Barad, Director of Clinical Research, Center for Human Reproduction
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09012010-01
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Infertility, Female
Keywords: Thin Endometrium; Asherman's Syndrome; Endometrial Scarring
MeSH Terms: conditions — Infertility, Female; Gynatresia | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (Experimental): G-CSF 300 units administered by trans-cervical infusion one time on day of hCG trigger for Ovulation
  Interventions: Drug: G-CSF
- Saline (Placebo Comparator): Saline administered by trans-cervical infusion one time on day of hCG trigger for ovulation
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: G-CSF — One infusion of G-CSF 300 units administered by intrauterine infusion
  Other Names: NEUPOGEN (Filgrastim)
  Arms: G-CSF
Drug: Saline — One intrauterine saline infusions of 1 cc
  Other Names: Normal Saline (Salt water); 0.91% w/v of NaCl, about 300 mOsm/L
  Arms: Saline

SUMMARY:
The purpose of this study is to investigate the effect of G-CSF on endometrial thickness in women who have failed reaching minimal endometrial thickness by standard treatments, to assess how many reach embryo transfer and what implantation and pregnancy rates are in comparison to control patients. The study will be conducted in women undergoing transfer of previously cryopreserved embryos or undergoing transfer of embryos from donor eggs.

DETAILED DESCRIPTION:
Objective: To investigate the effect of treatment with CSF : A placebo controlled double blinded crossover study.

Design: Crossover Randomized Control Trial

Setting: Academically affiliated private infertility centers

Subjects: Female IVF patients of all ages who are willing to be randomized to treatment and, in either IVF treatment, frozen embryo cycles (FET) or donor IVF cycles (D-IVF), 5 days before ET, have inadequate endometrial thickness.

Interventions: Subjects receive transvaginally, utilizing an insemination catheter, 2 slow intrauterine lavages with CSF-1 (Neupogen or generic, 300ug in 1 ml) 5 and 3 days, respectively, before embryo transfer and controls receive 1 ml of saline instead. Patients who do not become pregnant will after one month washout times continue treatment in the opposite study arm if they so choose and if they have remaining embryos.

Main Outcome Measures: Number of patients reaching embryo transfer with adequate endometrial thickness of at least 7mm.

Second Outcome Measures: Implantation and pregnancy rates..

Statistical and Power considerations: This is a Randomized Controlled Trial (RCT) with two study arms and panned crossover. Patients will be randomly assigned to Study group A or B according to a computer generated randomization table with 50:50 distributions. The study will test the null hypothesis that there is no difference in the transfer rates between the two groups. Transfer is only possible if the endometrial thickness reaches 7 mm or more. Order of treatment ab v ba will be added to the models as a separate factor and each phase will be analyzed as separate treatment strata.

The investigators are planning a study of independent cases and controls with 1 control per case. Prior data indicate that the transfer rate among controls is < 1%. If the true transfer rate for experimental subjects is 25%, the investigators will need to study 38 experimental subjects and 38 control subjects to be able to reject the null hypothesis that the transfer rates for experimental and control subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. We will use a continuity-corrected chi-squared statistic or Fisher's exact test to evaluate this null hypothesis.

There will be a planned interim analysis after 20 participants have completed the trial and if significant effects are observed the trial may be terminated at that time. The power to detect a difference in this interim analysis is only 42.6%.

ELIGIBILITY:
Inclusion Criteria:

* Patient's preparing for invitro fertilization and embryo transfer with endometrial growth of less than 7 mm, unresponsive to standard treatment

Exclusion Criteria:

* Sickle Cell disease
* Renal insufficiency
* Upper respiratory infection or Pneumonia
* Chronic Neutropenia
* Known Past or present malignancy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Barad, MD, MS, Principal Investigator — Center for Human Reproduction; Norbert Gleicher, MD, Study Chair — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients presenting for embryos transfer between October 3, 2010, and January 1, 2013, were offered participation in the trial. A total of 419 eligible patients were offered participation: Only 12 patients consented to participate in this study,(129 addtional patient participated in the NCT01202656 study) and 278 declined.
Pre-assignment Details: The principal reasons for refusal to participate were ''lack of interest'' and technical difficulties in presenting in timely fashion for the treatment to the center. Women with renal disease, sickle cell disease, or a history of malignancy were considered ineligible. No consenting patient was excluded from participation for medical reasons.
Groups:
- G-CSF Then Saline: G-CSF 300 units administered by trans-cervical infusion one time on day of hCG trigger for Ovulation then Saline administered by trans-cervical infusion one time on day of hCG trigger for ovulation
- Saline Then G-CSF: Saline administered by trans-cervical infusion one time on day of hCG trigger for ovulation then G-CSF 300 units administered by trans-cervical infusion one time on day of hCG trigger for Ovulation
Period: Period 1
Arm/Group | G-CSF Then Saline | Saline Then G-CSF
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Crossover Cycle
Arm/Group | G-CSF Then Saline | Saline Then G-CSF
Started (Patients were invited to the crossover but most chose not to continue in the study) | 1 (One patient became pregnant following Period 1, Only one non-pregnant chose to cycle again) | 2 (Three patients became pregnant after Period 1, 1 patient chose not to cycle again)
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The transfer rate among controls should be < 1%. If the true transfer rate for experimental subjects is 25%, we will need to study 38 experimental subjects and 38 control subjects to be able to reject the null hypothesis that the transfer rates for experimental and control subjects are equal with probability (power) 0.8.
Groups:
- Total: Total of all reporting groups
Arm/Group | G-CSF Then Saline | Saline Then G-CSF | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.79 (5.13) | 39.38 (6.03) | 39.59 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
FSH [Mean (Standard Deviation); unit: mIU/mL] — Day 3 Follicle Stimulating Hormone as a measure of baseline ovarian reserve
  mIU/mL | 8.64 (3.92) | 8.27 (4.01) | 8.46 (3.95)
Endometrial Thickness [Mean (Standard Deviation); unit: mm] | 5.6 (0.22) | 6.2 (0.69) | 5.8 (0.46)

OUTCOME MEASURES:

1. Primary Outcome: Endometrial Thickness
Description: Thickness of the endometrium on the day of embryo transfer
Time Frame: Day of embryo transfer
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | G-CSF | Saline
Number analyzed (Participants) | 8 | 7
mm | 11.3 (3.1) | 7.8 (0.8)
Statistical Analysis 1: Comparison: G-CSF vs Saline; Test type: Superiority or Other; p = 0.67, ANCOVA

2. Secondary Outcome: Implantation Rate
Description: Number of gestational sacs per number of embryos transferred in each treatment group
Time Frame: 28 days after embryo transfer
Population: Presuming an implantation rate of 10% and anticipating a 10% increase to 20% with treatment, about 200 embryos transferred in each study arm would be needed for 80% power and alpha of 0.05.
Measure: Number; unit: Gestational sacs
Units Other Than Participants: embryos transferred
Arm/Group | G-CSF | Saline
Number analyzed (Participants) | 8 | 7
Number analyzed (embryos transferred) | 14 | 18
Gestational sacs | 1 | 2
Statistical Analysis 1: Comparison: G-CSF vs Saline; Study was closed due to insufficient recruitment; Test type: Superiority or Other; p = 0.74, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | G-CSF | Saline
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No